CLINICAL TRIAL: NCT00988845
Title: Effects of Dietary Indole-3-Carbinol on Estrogen Metabolites Across a Wide Range of Body Mass Index: Implications for the Prevention of Endometrial Cancer in Obese Women
Brief Title: Indole-3-Carbinol Effects on Estrogen Metabolism
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual in the high BMI group
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: H-2009-0093; CC09709 (Other: UW Carbone Cancer Center); A532800 (Other: UW Madison); SMPH\OBSTET & GYNECOL\OB-GYN (Other: UW Madison)
Record Dates: First submitted 2009-10-01; First posted 2009-10-02 (Estimated); Last update posted 2019-12-13 (Actual); Status verified 2015-04

CONDITIONS: Obesity
Keywords: dietary supplement; indole 3 carbinol; estrogen
MeSH Terms: conditions — Obesity | interventions — indole-3-carbinol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Indole-3-carbinol (Experimental)
  Interventions: Dietary Supplement: Indole-3-carbinol

INTERVENTIONS:
Dietary Supplement: Indole-3-carbinol — 200 mg bid po X 8 weeks

SUMMARY:
This study will test a dietary supplement, indole-3-carbinol, for improving the estrogen profile in women across a range of body mass index.

ELIGIBILITY:
Inclusion Criteria:

* woman aged from 30 - 50 years
* regular menstrual cycle

Exclusion Criteria:

* taking hormone replacement or hormonal contraception
* thyroid disorder
* uncontrolled asthma
* BMI under 18.5
* allergy to cruciferous vegetables

Ages: 30 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2009-09; Primary Completion 2010-07 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Change in urinary 2/16-hydroxyestrone ratio | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Joseph P Connor, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States